CLINICAL TRIAL: NCT02123849
Title: The Effect of Intermittent Versus Continuous Dose Aspirin (ASA) on Nasal Epithelium Gene Expression in Current Smokers
Brief Title: Intermittent or Continuous Acetylsalicylic Acid and Gene Expression in the Nasal Tissue of Current Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2014-01006; NCI-2014-01006 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00031; HHSN2612012000311; 1300000502 (Other: The University of Arizona Medical Center-University Campus); UAZ2013-01-01 (Other: DCP); N01CN00031 (NIH); P30CA023074 (NIH)
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Results first posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Lung Carcinoma; Tobacco Use Disorder
MeSH Terms: conditions — Lung Neoplasms; Tobacco Use Disorder | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (continuous aspirin) (Experimental): Participants receive aspirin PO QD for 12 weeks.
  Interventions: Drug: Aspirin; Other: Laboratory Biomarker Analysis
- Arm II (intermittent aspirin) (Experimental): Participants receive placebo PO QD during weeks 1, 3, 5, 7, 9, and 11 and aspirin PO QD during weeks 2, 4, 6, 8, 10, and 12.
  Interventions: Drug: Aspirin; Other: Laboratory Biomarker Analysis; Other: Placebo

INTERVENTIONS:
Drug: Aspirin — Given PO
  Other Names: Acetylsalicylic Acid; ASA; Aspergum; Ecotrin; Empirin; Entericin; Extren; Measurin
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (intermittent aspirin)

SUMMARY:
This randomized phase II trial studies the safety and effects of acetylsalicylic acid (aspirin) taken continuously or intermittently on gene expression in the nasal tissue of current smokers. Smokers are at increased risk of developing lung cancer. Acetylsalicylic acid may be useful in preventing lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To analyze the impact of a 12-week intervention of intermittent and continuous acetylsalicylic acid (ASA) on a smoking-related gene expression signature in the nasal epithelium of current smokers and to analyze any difference between the intermittent and continuous ASA interventions.

SECONDARY OBJECTIVES:

I. To determine whether the change in the smoking-related gene expression signature of nasal epithelium persists one week off agent intervention.

II. To compare the change in urinary prostaglandin E metabolite (PGE-M) and leukotriene E (4) (LTE [4]) between the continuous and intermittent dosing arms and to determine whether the change persists one week off agent intervention.

III. To analyze the impact of intermittent and continuous ASA on a three lung cancer-related gene signatures (an 80-gene signature, a phosphoinositide 3-kinase [PI3K] gene signature, and a nasal epithelium cancer signature) in the nasal epithelium and to analyze any difference between the intermittent and continuous ASA interventions.

IV. To determine whether the change, if any, in the lung cancer-related gene expression signatures of nasal epithelium persists one week off agent intervention.

V. To compare the safety in current smokers of 12 week exposure to continuous versus intermittent ASA.

VI. To evaluate a gender effect in the modulatory effects of intermittent and continuous ASA on smoking-related gene expression signature.

VII. To explore in a discovery-driven fashion the effect of ASA intervention on whole-genome gene expression.

VIII. To analyze the impact of intermittent and continuous ASA on karyometric analysis of buccal cells and to analyze any difference between intermittent and continuous ASA interventions.

OUTLINE: Participants are randomized to 1 of 2 treatment arms.

ARM I (CONTINUOUS): Participants receive aspirin orally (PO) once daily (QD) for 12 weeks.

ARM II (INTERMITTENT): Participants receive placebo PO QD during weeks 1, 3, 5, 7, 9, and 11 and aspirin PO QD during weeks 2, 4, 6, 8, 10, and 12.

After completion of study treatment, participants are followed up for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female current tobacco smokers with >= 20 pack years of self-reported smoking exposure and an average use of >= 10 cigarettes/day
* Karnofsky >= 70%
* Leukocytes >= 3,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Hematocrit within normal institutional limits
* Platelets within normal institutional limits
* Total bilirubin =< 1.5 × institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 × institutional ULN
* Creatinine =< the upper institutional limits
* Prothrombin time (PT)/partial thromboplastin time (PTT) within normal institutional limits
* Fertile subjects must use adequate contraception (abstinence, barrier methods, or birth control pills) prior to study entry and for the duration of study participation
* Participants may have a history of indeterminate pulmonary nodule(s) by chest imaging if nodule follow-up has been completed or the study procedures would not interfere with nodule follow-up
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of allergic reaction to aspirin or attributed to compounds of similar chemical or biologic composition to aspirin, including other nonsteroidal anti-inflammatory drugs (NSAIDs)
* Gastric intolerance attributable to ASA or NSAIDs
* History of gastric ulcer within the past 5 years (with or without bleeding)
* Use of ASA or NSAIDs for more than 5 days per month within 3 months of enrollment
* Not willing or are unable to refrain from use of any non-study ASA or NSAIDs during the study period
* Adult asthma
* Chronic, current or recent (within the past three months) use of leukotriene antagonists
* Require chronic anticoagulation or anti-platelet therapy
* History of bleeding disorder or hemorrhagic stroke
* Chronic, current or recent (within the past three months) use of glucocorticoids (systemic, topical and/or nasal sprays)
* History of chronic sinusitis or recent nasal polyps
* Not willing or are unable to limit alcohol consumption to =< 2 alcoholic beverages a day during the study period
* Pregnant or lactating women; breastfeeding should be discontinued if the mother is treated with aspirin; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Participants may not be receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Have a known history of inability to absorb an oral agent
* Invasive cancer within the past five years except non-melanoma skin cancer
* Urine cotinine level, if collected at screening, does not confirm active smoking status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-06; Primary Completion 2016-09 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Garland, Principal Investigator — The University of Arizona Medical Center-University Campus
Locations (2):
- United States (2):
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Boston University School of Medicine, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Continuous Aspirin) | Arm II (Intermittent Aspirin)
Started | 27 | 27
Completed | 23 | 18
Not Completed | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Continuous Aspirin) | Arm II (Intermittent Aspirin) | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (8) | 52 (8) | 52 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 21 | 23 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 24 | 21 | 45
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Smoking-related Gene Expression Signature Score in Nasal Epithelium
Description: Change in nasal smoking-related gene expression signature score derived from prior research was compared between the two study arms. Prior research showed that a higher score was observed in never smokers compared to current smokers. An increased score implicated a more favorable intervention effect. There is no minimum or maximum score.
Time Frame: Baseline to 12 weeks (End-of-Intervention)
Population: The number of participants analyzed is different from the numbers provided in the Participant Flow Module because gene expression analysis was restricted to samples that met quality metrics.
Measure: Mean (Standard Deviation); unit: gene expression signature score
Arm/Group | Arm I (Continuous Aspirin) | Arm II (Intermittent Aspirin)
Number analyzed (Participants) | 22 | 14
gene expression signature score | -1.11 (4.05) | 1.39 (4.41)
Statistical Analysis 1: Comparison: Arm I (Continuous Aspirin) vs Arm II (Intermittent Aspirin); Test type: Non-Inferiority — The non-inferiority margin is 10% of the coefficient of variation (i.e., standard deviation divided by mean) which means that the changes in the signature score in the intermittent arm is no less than 90% of the coefficient of variation of the changes in the signature score in the continuous arm; p = 0.04, t-test, 1 sided

2. Secondary Outcome: Changes in Urine Leukotriene E4 (LTE(4)) Levels
Description: Urinary LTE(4) was used as a biomarker 5-lipoxygenase (5-LOX) mediated arachidonic acid metabolism. Decreased LTE4 implicated inhibition of the 5-LOX mediated pathway.
Time Frame: Baseline to 12 weeks (End-of-Intervention)
Measure: Mean (Standard Deviation); unit: pg/mg creatinine
Arm/Group | Arm I (Continuous Aspirin) | Arm II (Intermittent Aspirin)
Number analyzed (Participants) | 23 | 18
pg/mg creatinine | -6.89 (95.16) | -21.90 (309.8)
Statistical Analysis 1: Comparison: Arm I (Continuous Aspirin) vs Arm II (Intermittent Aspirin); Test type: Other; p = 0.84, t-test, 2 sided

3. Secondary Outcome: Changes in Urine Prostaglandin E2 Metabolite (PGE-M) Levels
Description: Urinary PGE-M was used as a biomarker of cyclooxygenase (COX) mediated arachidonic acid metabolism. Decreased PGE-M implicated inhibition of COX mediated pathway.
Time Frame: Baseline to 12 weeks (End-of-Intervention)
Measure: Mean (Standard Deviation); unit: ng/mg creatinine
Arm/Group | Arm I (Continuous Aspirin) | Arm II (Intermittent Aspirin)
Number analyzed (Participants) | 23 | 18
ng/mg creatinine | -3.73 (9.69) | -5.59 (13.74)
Statistical Analysis 1: Comparison: Arm I (Continuous Aspirin) vs Arm II (Intermittent Aspirin); Test type: Other; p = 0.61, t-test, 2 sided

4. Secondary Outcome: Number of Participants Experiencing Possibly/Probably/Definitely-related Adverse Events
Time Frame: Up to 2 weeks post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Continuous Aspirin) | Arm II (Intermittent Aspirin)
Number analyzed (Participants) | 27 | 27
Participants | 3 | 4
Statistical Analysis 1: Comparison: Arm I (Continuous Aspirin) vs Arm II (Intermittent Aspirin); Test type: Other; p = 1.00, Fisher Exact

5. Secondary Outcome: Gender Effect on Smoking-related Gene Expression Signature Score
Description: Change in nasal smoking-related gene expression signature score was compared between male and female participants. The gender comparison was not stratified by arm because of the small sample size. Prior research showed that a higher score was observed in never smokers compared to current smokers. An increased score implicated a more favorable intervention effect. There is no minimum or maximum score.
Time Frame: Baseline to 12 weeks (End-of-Intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gene expression signature score
Groups:
- Males (Overall): Male participants receive continuous or intermittent PO dosing of aspirin for 12 weeks.
- Females (Overall): Female participants receive continuous or intermittent PO dosing of aspirin for 12 weeks
Arm/Group | Males (Overall) | Females (Overall)
Number analyzed (Participants) | 18 | 18
gene expression signature score | 0.45 (5.04) | -0.72 (3.48)
Statistical Analysis 1: Comparison: Males (Overall) vs Females (Overall); Test type: Other; p = 0.42, t-test, 2 sided

6. Secondary Outcome: Changes in Lung Cancer-related Gene Expression Signature Score in the Nasal Epithelium
Description: Change in lung cancer-related gene expression signature score derived from prior research was compared between the two study arms. Prior research showed that the score was higher in lung cancer cases than healthy controls. A decreased score implicated a more favorable intervention effect. There is no minimum or maximum score.
Time Frame: Baseline to 12 weeks (End-of-Intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gene expression signature score
Arm/Group | Arm I (Continuous Aspirin) | Arm II (Intermittent Aspirin)
Number analyzed (Participants) | 22 | 14
gene expression signature score | -0.03 (0.12) | 0.04 (0.11)
Statistical Analysis 1: Comparison: Arm I (Continuous Aspirin) vs Arm II (Intermittent Aspirin); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.97, t-test, 1 sided

7. Secondary Outcome: Persistence of the Change in the Lung Cancer-related Gene Expression Signature Score in the Nasal Epithelium One Week Off Agent Intervention
Description: Change in the lung cancer-related gene expression signature score from baseline to one week off agent intervention was compared between the two study arms. Prior research showed that higher scores were observed in lung cancer cases than healthy controls. A decreased score implicated a favorable intervention effect. There is no minimum or maximum score.
Time Frame: Baseline to 1 week post-intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gene expression signature score
Arm/Group | Arm I (Continuous Aspirin) | Arm II (Intermittent Aspirin)
Number analyzed (Participants) | 21 | 14
gene expression signature score | -0.04 (0.09) | 0.02 (0.1)
Statistical Analysis 1: Comparison: Arm I (Continuous Aspirin) vs Arm II (Intermittent Aspirin); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.97, t-test, 1 sided

8. Secondary Outcome: Persistence of the Change in the Smoking-related Gene Expression Signature Score in the Nasal Epithelium One Week Off Agent Intervention
Description: Change in nasal smoking-related gene expression signature score from baseline to 1 week post-intervention was compared between the two study arms. Prior research showed that a higher score was observed in never smokers compared to current smokers. An increased score implicated a more favorable intervention effect. There is no minimum or maximum score.
Time Frame: Baseline to 1 week post-intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gene expression signature score
Arm/Group | Arm I (Continuous Aspirin) | Arm II (Intermittent Aspirin)
Number analyzed (Participants) | 21 | 14
gene expression signature score | -1.95 (3.42) | -0.1 (3.38)
Statistical Analysis 1: Comparison: Arm I (Continuous Aspirin) vs Arm II (Intermittent Aspirin); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.06, t-test, 1 sided

9. Secondary Outcome: Whole-genome Gene Expression - Number of Canonical Pathways Differentially Expressed
Description: Gene set enrichment analysis was performed on the MSigDB canonical pathways with the intent to discover differentially expressed genes after aspirin intervention.
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Number; unit: canonical pathway
Arm/Group | Arm I (Continuous Aspirin) | Arm II (Intermittent Aspirin)
Number analyzed (Participants) | 22 | 14
canonical pathway | 301 | 120

10. Secondary Outcome: Change in Buccal Cells Via Karyometric Analysis
Time Frame: Baseline to up to one week post-intervention
Population: Data were not collected
Arm/Group | Arm I (Continuous Aspirin) | Arm II (Intermittent Aspirin)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time that the first dose of study drug was taken until 2 weeks after participants come off the 12-week agent intervention.
Arm/Group | Arm I (Continuous Aspirin) | Arm II (Intermittent Aspirin)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 14/27 | 21/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Continuous Aspirin) (N=27) | Arm II (Intermittent Aspirin) (N=27)
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Upper Respiratory Infection (Injury, poisoning and procedural complications) | 2 | 4
Flu like syndromes (General disorders) | 1 | 2
Bruising (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 2
Injury, poisoning and procedural complications, others (Injury, poisoning and procedural complications) | 1 | 2
Weight gain (Investigations) | 4 | 3
Weight loss (Investigations) | 0 | 5
Dizziness (Nervous system disorders) | 0 | 2
Headache (Pregnancy, puerperium and perinatal conditions) | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less